CLINICAL TRIAL: NCT04553601
Title: Molecular Imaging Visualization of Tumor Heterogeneity in Non-small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KYH2019-039
Record Dates: First submitted 2020-07-30; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-07

CONDITIONS: NSCLC; PET/CT; Biopsy; Radiomics; Genomics; Whole-exome Sequencing
Keywords: NSCLC, PET/CT, radiogenomics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Patients with advanced NSCLC underwent 18F-FDG PET/CT and PET/CT-guided synchronous targeted biopsy of primary and distant metastatic tumors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 8F-FDG PET/CT and PET/CT-guide targeted biopsy (Experimental): Each subject receive a single intravenous injection of 18F-FDG PET/CT and PET/CT-guide targeted biopsy within the specified time.
  Interventions: Diagnostic Test: 18F-FDG PET/CT and PET/CT-guide targeted biopsy in another group of participants

INTERVENTIONS:
Diagnostic Test: 18F-FDG PET/CT and PET/CT-guide targeted biopsy in another group of participants — Each subject receive a single intravenous injection of 18F-FDG PET/CT and PET/CT-guide targeted biopsy within the specified time

SUMMARY:
To assess the potential usefulness of radiogenomics for tumor driving genes heterogeneity in non-small cell lung cancer.

DETAILED DESCRIPTION:
Patients with advanced NSCLC underwent 18F-FDG PET/CT and PET/CT-guided synchronous targeted biopsy of primary and distant metastatic tumors. The LIFEx package was used to extract PET and CT radiomic features from primary and metastatic lesions. The radiomic ROI sites of primary and distant metastatic tumors were point-to-point corresponding to the PET/ CT-guided targeted biopsy sites. Whole exon sequencing of primary and distant metastatic tumor samples obtained by PET/CT-guided targeted biopsy was used to get genomic data of primary and distant metastatic tumor. Predictive radiogenomics models were established and validation.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* (i) adult patients (aged 18 years or order);
* (ii) patients with suspected or newly diagnosed or previously treated malignant tumors (supporting evidence may include magnetic resonance imaging (MRI), CT, tumor markers and pathology report);
* (iii) patients who had scheduled both 18F-FDG PET/CT scans and PET/CT guided biopsy;
* (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* (i) patients with non-malignant lesions;
* (ii) patients with pregnancy;
* (iii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Radiomic feature selection and model establishment | 3 years
  In this study, the investigators first selected the features with significant differences between genes mutant and wild type in the training set using the Mann-Whitney U test, obtaining a total of 53 features with p value < 0.05. Then, the least absolute shrinkage and selection operator (LASSO) algorithm was used to select the optimal predictive features among the 53 selected in the training set. The LASSO algorithm adds a L1 regularization term to a least square algorithm to avoid overfitting. A prediction model was established by logistic regression, and the radiomics signature score (rad-score) for each participant was calculated based on the selected discriminating radiomic features. The model performance was tested in the validation set. The receiver operating characteristic (ROC) curve and the area under the curve (AUC) were used to evaluate the model performance in the training and validation sets.

SECONDARY OUTCOMES:
Genes mutation detection | 30 days
  Genes mutation detection was performed on histological specimens obtained by surgical resection or puncture. Genes mutation detection was conducted by the examination of the whole-exome sequencing. The whole-exome sequencing is performed by the Novogene company (www.novogene.com). If any genes mutation in the whole-exome sequencing was detected, the tumor was considered genes mutant. Otherwise, the tumor was classified as no mutant of genes type.
Image acquisition | 30 days
  The imaging acquisition protocol was established following the Image Biomarker Standardisation Initiative (IBSI) reporting guidelines. All the details of the procedures are provided in the electronic supplementary material. 18F-FDG PET/CT (Discovery MI, GE Healthcare, Milwaukee, WI, USA) examination was performed within 1 month before treatment. Briefly, 18F-FDG PET/CT images were acquired 60 ± 5 min after 18F-FDG injection in accordance with the European Association of Nuclear Medicine (EANM) guidelines, version 1.0 (version 2.0 from February 2015). A 3D LOR reconstruction algorithm was used to reconstruct the PET images. The attenuation correction of PET images was carried out with CT data, and the corrected PET images were fused with CT images.
Radiomic feature extraction | 30 days
  The LIFEx package (version 4.00, http://www.lifexsoft.org) was used to extract the texture features of PET/CT images of lesions in the same VOI. The PET/CT image of the patient in the DICOM format was imported into the software. Two experienced PET/CT diagnostic physicians semi-automatically delineated the region of interest of the target lesion using a threshold of 40% of the maximum standardized uptake value (SUVmax). Then, the software program automatically calculates and extracts 47 PET radiomic features and 45 CT radiomic features.

CONTACTS AND LOCATIONS:
Overall Officials: Long Sun, PhD, Principal Investigator — The First Affiliated Hospital of Xiamen University
Locations (1):
- First affiliated hospital of xiamen university, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No